CLINICAL TRIAL: NCT02002273
Title: The Effect of Regulated Pleural Pressure on The Duration of Air Leak and Fluid Drainage Following Pulmonary Anatomic Resections: A Multicenter Randomized Trial
Brief Title: Effect of Regulated Pleural Pressure on Air Leak and Fluid Drainage Following Pulmonary Resections: A Multicenter Randomized Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedali Riuniti Ancona (Other)
Collaborators: The Leeds Teaching Hospitals NHS Trust (Other); Yale University (Other); The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cecilia Pompili, MD, Ospedali Riuniti Ancona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Airleak-2013-1
Record Dates: First submitted 2013-11-29; First posted 2013-12-05 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

ARMS (2):
- Patients with regulated suction mode (Experimental): On the morning of each postoperative day (starting with POD#1) patients of group 1 are switched for 4 hours to -8 cm H2O After this period of 4 hours both groups are switched back to their original pressure levels, with the effect on air leak and fluid leak measured. Pts are then left on their original pressure level until the next day, when the switch to -8 or - 20 cm H2O is again made.
  Interventions: Procedure: Switching level of suction
- regulated seal mode (-8 cmH2O). (Experimental): On the morning of each postoperative day (starting with POD#1) patients of group 1 are switched for 4 hours to -8 cm H2O and patients of group 2 are switched to -20 cm H2O. After this period of 4 hours both groups are switched back to their original pressure levels, with the effect on air leak and fluid leak measured. Pts are then left on their original pressure level until the next day, when the switch to -8 or - 20 cm H2O is again made.
  Interventions: Procedure: Switching level of suction

INTERVENTIONS:
Procedure: Switching level of suction

SUMMARY:
The objective of this randomized study is to compare the effect of two controlled chest tube protocols on the duration of air leak and fluid drainage following pulmonary lobectomy or segmentectomy by using an electronic regulated chest drainage system (Thopaz). Previous studies have suggested that the amount of negative pressure used at the level of the chest drainage device may affect the duration of air leak, but the results have been inconsistent, however as revealed in more recent studies understanding of the physics of chest drainage devices may have been confounded by lack of regulation of the pleural pressure.

In addition, experimental studies have shown that fluid drainage may be affected by the degree of negative pleural pressure applied.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to read, understand, and provide written Informed Consent;
* Age range of 18-90 years;
* Patients submitted to lobectomy, segmentectomy and bilobectomy due to lung cancer or other intrathoracic lesions. Both open and minimally invasive (thoracoscopic) resections are acceptable.

Exclusion Criteria:

* if patients are submitted to lung resection associated with chest wall resection or diaphragm resection the patient will be excluded from analysis
* If during the postoperative hospital course there is a need for postoperative mechanical ventilation or hemodynamic instability the patient will be excluded from analysis.
* If the subject meets all of the inclusion criteria and none of the exclusion criteria, he/she is eligible to participate in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
duration of air leak | up to 7 days

SECONDARY OUTCOMES:
1. Differences in airflow detected during the 4 hours after the pressure level is switched to -8 cmH2O or -20 cmH2O compared to the original pressure level in both groups | up to 5 days
Differences in fluid drainage | up to 5 days
Duration of chest tube left in the patient (days) | up to 7 days
Postoperative length of hospital stay (days) | up to 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedali Riuniti Ancona, Ancona, Italy